CLINICAL TRIAL: NCT07185243
Title: A Study Evaluating the Safety and Efficacy of hV01, a Recombinant Human IL-21-expressing Oncolytic Vaccinia Virus, in Combination With the PD-1 Inhibitor Tislelizumab for Advanced Solid Tumors.
Brief Title: A Study to Evaluate Combination Therapy of Oncolytic Vaccinia Virus (hV01) and PD-1 Inhibitor in Advanced Solid Tumors.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Converd Co., Ltd. (Industry)
Collaborators: Xiamen Humanity Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hV01-IST-02
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hV01 as a single agent, and combined with Tislelizumab (Experimental): Part A:
  The first group of participants will receive an intratumoral injection of hV01 on days 1 and 3 of each 28-day cycle.
  The second group of participants will receive an intratumoral injection of hV01 on days 1, 3, and 5 of each 28-day cycle.
  Part B:
  Based on the results from Part A, participants will receive an intratumoral injection of hV01 on days 1 and 3 or on days 1, 3, and 5, followed by intravenous infusion of Tislelizumab on days 14 and 35 of each 42-day cycle.
  Interventions: Biological: recombinant human IL-21-expressing oncolytic vaccinia virus injection

INTERVENTIONS:
Biological: recombinant human IL-21-expressing oncolytic vaccinia virus injection — hV01 is a recombinant vaccinia virus with deletions of the viral thymidine kinase (TK) and viral growth factor (VGF) genes and insertion of the human IL-21 gene.
  Other Names: hV01

SUMMARY:
The purpose of this study is to evaluate the safety and primary efficacy of the combination therapy of recombinant human IL-21-expressing oncolytic vaccinia virus (hV01) and the PD-1 Inhibitor Tislelizumab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is divided into two parts and follows a single-arm design.

Part A evaluates the safety and tolerability of hV01 administration at two different frequencies: twice per 28-day cycle (on days 1 and 3) and three times per 28-day cycle (on days 1, 3, and 5). The study will adhere to the 3+3 principle for monitoring dose-limiting toxicity (DLT).

Part B assesses the combination of hV01 and Tislelizumab. This phase will involve multiple administrations of hV01 (either twice or three times per 42-day cycle), followed by the administration of Tislelizumab on days 14 and 35. Monitoring for DLTs will also be conducted for the first 3 or 6 subjects in this phase.

Efficacy will be evaluated using the RECIST v1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signing an informed consent form.
2. Men or women aged 18 to 75 years.
3. Histologically and/or cytologically confirmed advanced solid tumors refractory or failed to respond to standard therapies.
4. At least one measurable lesion according to RECIST v1.1 criteria, which is suitable for intratumoral injection of hV01 either directly or with the assistance of B-ultrasound, or CT scan. The baseline longest diameter of the lesion targeted for injection should be more than 1.5 cm.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Life expectancy of at least 6 months.
7. Required baseline laboratory data include: (1) Hematology: absolute neutrophil count (ANC) ≥ 1.5×10^9/L, platelet (PLT) count ≥ 75×10^9/L, hemoglobin (Hb) ≥90 g/L; (2) Liver function: serum total bilirubin (TBIL) ≤1.5×ULN (or ≤3×ULN for patients with Gilbert's syndrome or liver metastasis); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3×ULN (or<5×ULN for patients with primary liver cancer or liver metastasis); (3) Renal function: serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance (Cockcroft-Gault method) ≥45 mL/min. For men: creatinine clearance = [[140-age(yr)]×weight (kg)]/[0.818×creatinine (μmol/L)]; For women: creatinine clearance = [[140-age(yr)]×weight (kg)×0.85]/[0.818×creatinine (μmol/L)]; (4) Coagulation test: activated partial thromboplastin time (APTT) ≤1.5×ULN; international normalized ratio (INR)≤1.5×ULN.
8. Female patients of childbearing age must have a negative serum pregnancy test. Note: non-childbearing potential as defined by at least one of the following criteria: surgeries resulted in permanent sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or are post-menopausal; For females aged 50 or older, they will be considered menopausal if they are in amenorrhea, defined as the absence of menstruation for the previous 12 months before screening, which is not caused by any disease; For females younger than 50 years, they will be considered menopausal if they satisfy all the following requirements during screening: they are in amenorrhea, defined as the absence of menstruation for the previous 12 months after termination of hormone treatment, and they have a serum FSH level within the laboratory's reference range for postmenopausal females.

Exclusion Criteria:

1. Receiving any of the following anti-tumor treatments within a specified time period: (1) Systemic anti-tumor treatment, including chemotherapy, large-molecule targeted therapy, immunotherapy, and endocrine therapy within 4 weeks before first dose of hV01 (within 6 weeks of dosing for nitrosourea or mitomycin C); (2) Small-molecule targeted therapy within 2 weeks before first dose of hV01 or within five half-lives of the small-molecule targeted drug (whichever is longer); (3)Radiotherapy (excluding palliative radiotherapy) within 2 weeks before first dose of hV01. (4) previous treatment with an oncolytic virus.
2. Receiving any investigational drugs for clinical trials within 4 weeks prior to the first dose of hV01.
3. Patients with clinical symptoms of central nervous system (CNS) metastasis or meningeal metastasis, or other evidence indicating that CNS or meningeal metastases are not controlled.
4. Known or suspected active autoimmune diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, and Hashimoto's thyroiditis).
5. Patients who have received an allogeneic stem cell transplant or organ transplant.
6. Patients with a history of severe cardiovascular and cerebrovascular diseases, including: (1) Acute coronary syndrome (including myocardial infarction, severe or unstable angina), myocarditis, congestive heart failure, cerebrovascular accidents, or other cardiovascular events of CTCAE (v5.0) grade 3 or higher within 12 months of first hV01 dosing; (2) Severe arrhythmia requiring clinical intervention; (3) New York Heart Association (NYHA) classification of class II or above, or left ventricular ejection fraction (LVEF) <50%; (4) Uncontrolled hypertension or hypotension despite standard treatment.
7. Clinically significant and/or rapidly accumulating pericardial and/or pleural effusion.
8. Bleeding symptoms of great clinical significance or clear bleeding tendency within six months prior to the initial dose of hV01.
9. Severe inflammatory skin diseases that require treatment with medicines (e.g., eczema or psoriasis requiring systematic treatment).
10. Any uncontrolled active infection requiring systemic anti-infective therapy (graded 2 or higher according to CTCAE v5.0), including but not limited to active tuberculosis, sepsis, bacteremia, fungemia, and viremia.
11. Any of the following infections: human immunodeficiency virus (HIV), syphilis spirochete(TP), active hepatitis C (positive HCV RNA test), or active hepatitis B (positive HBsAg and HBV DNA ≥ 2000 IU/mL or ≥10^4 copies/mL).
12. Receiving therapeutic dosages of corticosteroids such as prednisone or its equivalent >10 mg daily within two weeks prior to the first dose of hV01, or having any coexisting diseases that might require systemic corticosteroids or any other immune suppressors during the study (assessed by the investigators) with the following exceptions: local administration of glucocorticoid (e.g. topical routes such as for eyes, intra-articular, intranasal, or inhaled); or usage of glucocorticoids for a short period of time for preventive purposes such as for the prevention of contrast media hypersensitivity).
13. Receiving any of the live vaccines within four weeks of the first dose of hV01.
14. Patients with a history of severe allergies.
15. Mental disorders that could potentially impact the participant's ability to comply with the study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities | From the first hV01 dose till the end of cycle 1 (each cycle is 28 days in Part A and 42 days in Part B of the study).
  To observe dose-limiting toxicities (DLTs) after hV01 administration as a single agent, or combined with Tislelizumab.
Adverse events | From informed consent to approximately 3 months after the End of Treatment (EOT).
  Assess the frequency, severity, and nature of adverse events (AEs).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Until the first documented disease progression or death from any cause, up to 2 years after EOT.
  The proportion of patients who have a partial or complete response to therapy.
Disease Control Rate (DCR) | Until the first documented disease progression or death from any cause, up to 2 years after EOT.
  The percentage of participants who gain a complete response, a partial response, or stable disease.
Duration of Response (DOR) | Until the first documented disease progression or death from any cause, up to 2 years after EOT.
  The time from administration of the first dose of hV01 to disease progression or death in patients who achieve a complete or partial response.
Progression-Free Survival (PFS) | Until the first documented disease progression or death from any cause, up to 2 years after EOT.
  The time from administration of the first dose of hV01 to disease progression or death from any cause.
Overall Survival (OS) | Until the date of death from any cause, up to 2 years after EOT.
  The length of time from administration of the first dose of hV01 during which patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Huang, Principal Investigator — Xiamen Humanity Hospital
Locations (1):
- Xiamen Humanity Hospital, Xiamen, Fujian, China